CLINICAL TRIAL: NCT06862778
Title: Clinical Diagnosis of Diabetes Using Surface-enhanced Raman Spectroscopy Liquid Biopsy and Machine Learning
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Aachen (Other)
Collaborators: University of Agriculture Faisalabad (Unknown); Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Roger Molto Pallares, Group Leader, University Hospital, Aachen
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Diabetes SERS 01
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
Keywords: Diabetes; Sensing; SERS; Gold nanoparticles; Diagnositcs; Surface-enhanced Raman Spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Experimental): The Raman spectra of healthy patient samples will be measured in the presence of gold nanoparticles, which will enhance the spectroscopic characteristics of serum components via near-field enhancements.
  Interventions: Diagnostic Test: SERS
- Diabetes (Experimental): The Raman spectra of diabetic patient samples will be measured in the presence of gold nanoparticles, which will enhance the spectroscopic characteristics of serum components via near-field enhancements.
  Interventions: Diagnostic Test: SERS

INTERVENTIONS:
Diagnostic Test: SERS — Spectroscopic assessment of serum samples from healthy and diabetic patients to identify characteristics for diagnosis.
  Other Names: Surface-enhanced Raman Spectroscopy

SUMMARY:
This project aims to adapt the gold nanoparticle-based surface-enhanced Raman spectroscopy (SERS) technology to clinical application. In this exploratory study, a measurement protocol will be established to investigate whether SERS (combined with multivariate data analysis or machine learning algorithms) allows the diagnosis of patients with diabetes.

DETAILED DESCRIPTION:
This study on the clinical application of surface-enhanced Raman spectroscopy (SERS) comprises two parts. First, a SERS measurement protocol will be developed to enhance the interactions between gold nanoparticles and the components of the patient's samples, maximizing Raman spectroscopical signatures. Given the complex composition of human blood, which encompasses numerous biological constituents, the study focuses on serum, a component obtained through centrifugation after removing cells and clotting factors. Fifteen spectra will be recorded per sample. The raw spectra will be post-processed, including removal of the substrate signal, baseline correction, vector normalization, and smoothing steps.

The SERS measurement protocol established in the first section will subsequently be applied to samples of healthy and diabetes patients. Two different approaches will be followed. First, multivariate data analysis will be performed to identify distinctive feature characteristics in the samples that correlate to their group (healthy and diabetes patients), allowing patient diagnosis. Second, different machine learning algorithms and data augmentation strategies will be explored for better patient diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Nishtar Medical University
* Patient age from 18 to 70 years
* Confirmed disease (for diabetic group)

Exclusion Criteria:

* Patients with severe concurrent diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
SERS measurements to differentiate between healthy and diabetic patients | Through study competition, up to 1 year
  SERS assessment of healthy and diabetic patient samples to identify unique spectroscopical characteristics to discriminate between healthy and diabetic patients

CONTACTS AND LOCATIONS:
Locations (1):
- RWTH Aachen university hospital, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided